CLINICAL TRIAL: NCT01069003
Title: EDUCATE: a Prospective, Multi-center Study Designed to Collect Real-world Safety and Clinical Outcomes in Subjects Receiving One or More Endeavor Zotarolimus-Eluting Stents and Either Clopidogrel and Aspirin or Prasugrel and Aspirin as Part of a Dual Antiplatelet Therapy (DAPT) Drug Regimen
Brief Title: EDUCATE: The MEDTRONIC Endeavor Drug Eluting Stenting: Understanding Care, Antiplatelet Agents and Thrombotic Events
Acronym: EDUCATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IP114
Record Dates: First submitted 2010-02-12; First posted 2010-02-17 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: Heart Disease; Cardiovascular Disease; Platelet Aggregation Inhibitors; Dual Antiplatelet Therapy; Clopidogrel; Prasugrel; Vascular Disease; Myocardial Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Arm (Placebo Comparator): Subjects are randomized to receive 18 months of placebo thienopyridine and aspirin (ASA). Eligible subjects are without death, myocardial ischemia, stroke, repeat coronary revascularization, major bleeding or stent thrombosis in the first 12 months prior to randomization.
  Interventions: Drug: Placebo Arm
- Thienopyridine Therapy (Active Comparator): Subjects are randomized to receive 18 months of active thienopyridine and aspirin (ASA). Eligible subjects are without death, myocardial ischemia, stroke, repeat coronary revascularization, major bleeding or stent thrombosis in the first 12 months prior to randomization.
  Interventions: Drug: Thienopyridine Therapy
- Surveillance Arm (Other): Non randomized subjects followed through 24 months
  Interventions: Device: Surveillance Arm

INTERVENTIONS:
Drug: Placebo Arm — Placebo and ASA (75 mg - 325 mg)
  Arms: Placebo Arm
Drug: Thienopyridine Therapy — Prasugrel 5 or 10 mg or Clopidogrel 75 mg plus ASA (75 mg - 325 mg)
  Arms: Thienopyridine Therapy
Device: Surveillance Arm — Non randomized arm to understand clinical outcomes in a commercial setting
  Arms: Surveillance Arm

SUMMARY:
EDUCATE is a prospective, multi-center study designed to collect real-world safety and clinical outcomes in subjects receiving one or more Endeavor Zotarolimus-Eluting Stents and either clopidogrel and aspirin or prasugrel and aspirin as part of a dual antiplatelet therapy (DAPT) drug regimen.

DETAILED DESCRIPTION:
To provide clinical information on rates of late and very late stent thrombosis after Endeavor Drug-eluting Stent (DES)placement in an all comers population with a broad range of bleeding and thrombosis risk. EDUCATE will further analyze the current practice of clinicians regarding temporary cessation of antiplatelet therapy and its association with clinical outcomes. In addition, patients included in this broad Endeavor registry will also be contributed to the DAPT native study population for analysis of 12 vs 30 months duration of dual antiplatelet therapy.

ELIGIBILITY:
ENROLLMENT INCLUSION CRITERIA

* Patient is older than 18 years.
* The patient or patient's legal representative has consented to participate and has authorized the collection and release of his medical information by signing the "Subject Informed Consent Form".
* Patients undergoing percutaneous intervention with Endeavor stent deployment (or has within 24 hours).
* The patient is willing and able to cooperate with study procedures and required follow up visits.

ENROLLMENT EXCLUSION CRITERIA

* Index procedure stent placement with stent diameter < 2.5 mm or > 3.5 mm.
* Pregnant women.
* Current medical condition with a life expectancy of less than 3 years.
* The patient is currently participating in another investigational device or drug study that clinically interferes with the EDUCATE Study. The patient may only be enrolled in the EDUCATE Study once.
* Patients with hypersensitivity or allergies to one of the drugs or components indicated in the Instructions for Use.
* Patients in whom anti-platelet and/or anticoagulation therapy is contraindicated.
* Patients treated with any stent other than the Endeavor stent during the index procedure.

RANDOMIZATION INCLUSION CRITERIA AT 12 MONTHS

* Subject is "12 Month Clear".
* Subjects without known contraindication to dual antiplatelet therapy for at least 18 months after randomization.

RANDOMIZATION EXCLUSION CRITERIA AT 12 MONTHS

* Pregnant women.
* Subject switched thienopyridine type or dose within 6 months prior to randomization.
* Planned surgery necessitating discontinuation of antiplatelet therapy within the 18 months following randomization.
* Percutaneous coronary intervention or cardiac surgery between 6 weeks post index procedure and randomization.
* Planned surgery necessitating discontinuation of antiplatelet therapy within the 21 months following randomization.
* Current medical condition with a life expectancy of less than 3 years.
* Subjects on warfarin or similar anticoagulant therapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2272 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Cutlip, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Harold Dauerman, MD, Principal Investigator — Fletcher Allen Hospital
Locations (1):
- AnMed Health Medical Center, Anderson, South Carolina, United States

REFERENCES:
- [Derived] Cutlip DE, Kereiakes DJ, Mauri L, Stoler R, Dauerman HL; EDUCATE Investigators. Thrombotic complications associated with early and late nonadherence to dual antiplatelet therapy. JACC Cardiovasc Interv. 2015 Mar;8(3):404-410. doi: 10.1016/j.jcin.2014.10.017. Epub 2015 Feb 18. PMID 25703885
- See also: Native DAPT Study Web Site — http://www.daptstudy.org/
- See also: Harvard Clinical Research Institute — http://www.hcri.harvard.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled 2272 but only 2262 subjects were analysis receiving the Endeavor stent only.
Groups:
- Placebo: Subjects without death, MI, stroke, repeat coronary revascularization, major bleeding or stent thrombosis in the first 12 months. These subjects are randomized to receive 18 months of placebo thienopyridine and aspirin (ASA).
  Placebo (12-Month Arm): Placebo
  ASA: 75 mg - 325 mg Aspirin(ASA)
- Thienopyridine Therapy: Subjects without death, MI, stroke, repeat coronary revascularization, major bleeding or stent thrombosis in the first 12 months. These subjects are randomized to receive 18 months of active thienopyridine and aspirin (ASA).
  Prasugrel and Clopidogrel (30-Month Arm): Prasugrel 5 or 10 mg; Clopidogrel 75 mg
  ASA: 75 mg - 325 mg Aspirin(ASA)
- Surveillance Arm: Non randomized subjects followed for total of 24 months
Period: Overall Study
Arm/Group | Placebo | Thienopyridine Therapy | Surveillance Arm
Started | 399 | 412 | 1451
Completed | 353 | 358 | 976
Not Completed | 46 | 54 | 475

BASELINE CHARACTERISTICS:
Population: The intent to treat arm contains non randomized subjects followed through 24 months
Groups:
- Placebo Arm: Subjects without death, MI, stroke, repeat coronary revascularization, major bleeding or stent thrombosis in the first 12 months. These subjects are randomized to receive 18 months of placebo thienopyridine and aspirin (ASA).
  Placebo (12-Month Arm): Placebo
  ASA: 75 mg - 325 mg Aspirin(ASA)
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Thienopyridine Therapy | Surveillance Arm | Total
Number analyzed (Participants) | 399 | 412 | 1451 | 2262
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.7) | 62.5 (10.7) | 64.6 (11.3) | 63.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 116 | 449 | 687
  Male | 277 | 296 | 1002 | 1575
Region of Enrollment [Number; unit: participants]
  United States | 372 | 385 | 1409 | 2166
  Canada | 27 | 27 | 42 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite of All Death, Target Vessel Myocardial Infarction (MI) and Stroke (Defined as MACCE) for Randomized Subjects
Time Frame: Placebo and Thienopyridine 12 - 30 months; Surveillance Arm (0 - 24 months)
Measure: Number; unit: Percentage of participants
Groups:
- Surveillance Arm: Subjects followed for total of 24 months and not clear for randomization. Subjects who had a death, MI, stroke, repeat coronary revascularization, major bleeding or stent thrombosis in the first 12 months prior to randomization.
Arm/Group | Placebo Arm | Thienopyridine Therapy | Surveillance Arm
Number analyzed (Participants) | 392 | 393 | 1451
Percentage of participants | 4.3 | 4.8 | 16.9

2. Primary Outcome: Percentage of Participants of Incidence of ARC Definite or Probable Stent Thrombosis (ST) for Randomized Subjects
Description: All definite and probable Stent Thrombosis (ST) are adjudicated by an independent committee according to the definition based on Academic Research Consortium (ARC)
  Definite is defined as angiographic or pathologic confirmation of partial or total thrombotic occlusion within the peri-stent region and at least 1 of the following: Acute ischemic symptoms, Ischemic ECG changes, Elevated cardiac biomarkers
  Probable defined as any unexplained death within the first 30 days of procedure and any myocardial infarction, which is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause
Time Frame: Placebo and Thienopyridine 12 - 30 months; Surveillance Arm (0 - 24 months)
Measure: Number; unit: percentage of participants
Groups:
- Placebo Arm: Subjects without death, myocardial ischemia, stroke, repeat coronary revascularization, major bleeding or stent thrombosis in the first 12 months. These subjects are randomized to receive 18 months of placebo thienopyridine and aspirin (ASA).
  Placebo (12-Month Arm): Placebo
  ASA: 75 mg - 325 mg Aspirin(ASA)
- Thienopyridine Therapy: Subjects without death, myocardial ischemia, stroke, repeat coronary revascularization, major bleeding or stent thrombosis in the first 12 months. These subjects are randomized to receive 18 months of active thienopyridine and aspirin (ASA).
  Prasugrel and Clopidogrel (30-Month Arm): Prasugrel 5 or 10 mg; Clopidogrel 75 mg
  ASA: 75 mg - 325 mg Aspirin(ASA)
Arm/Group | Placebo Arm | Thienopyridine Therapy | Surveillance Arm
Number analyzed (Participants) | 392 | 393 | 1451
percentage of participants | 1.0 | 0.5 | 2.4

3. Primary Outcome: Incidence of Major Bleeding (GUSTO Classification, Severe and Moderate Bleeding Combined) for Randomized Subjects
Time Frame: Placebo and Thienopyridine 12 - 30 months; Surveillance Arm (0 - 24 months)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Arm | Thienopyridine Therapy | Surveillance Arm
Number analyzed (Participants) | 392 | 393 | 1451
Percentage of participants | 1.8 | 2.0 | 4.8

ADVERSE EVENTS:
Time Frame: All events were collected up to 12 months post procedure and only serous adverse events were collected after 12 months
Arm/Group | Placebo Arm | Thienopyridine Therapy | Surveillance Arm
Serious Adverse Events (participants affected / at risk) | 117/399 | 111/412 | 664/1451
Other Adverse Events (participants affected / at risk) | 0/399 | 0/412 | 90/1451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=399) | Thienopyridine Therapy (N=412) | Surveillance Arm (N=1451)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 15 (21)
Acute Myocardial Infarction (Cardiac disorders) | 7 (7) | 3 (3) | 55 (59)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 2 (2) | 37 (41)
Angina Pectoris (Cardiac disorders) | 10 (10) | 3 (3) | 39 (40)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0) | 31 (32)
Atrial Fibrillation (Cardiac disorders) | 6 (7) | 4 (4) | 24 (26)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4) | 9 (10)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 14 (14)
Cardiac Enzymes Increased (Investigations) | 0 (0) | 1 (1) | 15 (16)
Cardiac Failure Congestive (Cardiac disorders) | 3 (7) | 3 (3) | 39 (53)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1) | 3 (4)
Cerebrovascular Accident (Nervous system disorders) | 4 (4) | 3 (3) | 19 (22)
Chest Discomfort (General disorders) | 2 (2) | 2 (2) | 6 (6)
Chest Pain (General disorders) | 11 (12) | 9 (10) | 97 (128)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 20 (33)
Coronary Artery Disease (Cardiac disorders) | 13 (13) | 18 (20) | 0 (0)
Coronary Artery Occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 8 (8)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 4 (4) | 19 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 7 (7)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 5 (5) | 7 (7) | 44 (51)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 6 (6)
Haemorrhage (Vascular disorders) | 0 (0) | 2 (2) | 7 (8)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 12 (12)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 10 (11)
In-Stent Coronary Artery Restenosis (Cardiac disorders) | 3 (3) | 6 (6) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 3 (4) | 11 (13)
Myocardial Infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 3 (3) | 5 (7) | 15 (16)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 4 (4)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2) | 20 (26)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 7 (9)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4)
Renal Failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 14 (16)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Therapeutic Embolisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 2 (2)
Thrombosis In Device (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 18 (18)
Transient Ischaemic Attack (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 7 (9)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=399) | Thienopyridine Therapy (N=412) | Surveillance Arm (N=1451)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 90 (96)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other